CLINICAL TRIAL: NCT03230981
Title: Age-dependency of Cornea Biomechanics Measured by OCT Vibrography: A Pilot Study
Brief Title: Age-dependency of Cornea Biomechanics Using OCT Vibrography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Seok Hyun Yun, Professor of Dermatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017P000867
Record Dates: First submitted 2017-07-16; First posted 2017-07-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Cornea
Keywords: biomechanics; cornea; optical coherence tomography; vibrography; brillouin microscopy
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Optical imaging of the cornea in healthy subjects
  Interventions: Device: Optical imaging of the cornea in healthy subjects

INTERVENTIONS:
Device: Optical imaging of the cornea in healthy subjects — OCT vibrography and Brillouin microscopy

SUMMARY:
The aim of this pilot study is to assess the ability of a new optical coherence tomography system to obtain information on biomechanics of the cornea.

DETAILED DESCRIPTION:
The cornea, the clear front window of the eye, consists of finely intertwined collagen fibers, which give the cornea a microstructure that provides mechanical integrity necessary to maintain its typical dome-shape against the intraocular pressure (IOP). Changes in the biomechanical properties can lead to an abnormal corneal shape and refractive errors. As a result, light is not perfectly focused onto the retina and the vision is affected. A typical example of alterations in the cornea's biomechanical properties is found in patients with an eye disorder called Keratoconus, which leads to progressive thinning of the cornea. Numerous studies have shown that promising interventions like collagen crosslinking (CXL) can slow down an arrest progression of ectatic eye diseases. Keratoconus, as a typical example, although it cannot be cured, could be at least halted by CXL. Therefore, early diagnosis of ectasia is crucial for the patient. Current diagnostic methods of ectasia are based on morphological rather than biomechanical analysis. The irregular patterns of the cornea can be detected by pachymetry and topography before clinical signs occur, but these tests cannot reliably differentiate truly weak or keratoconic corneas from atypical normal ones.

These are compelling needs for improved diagnostic methods. More recently, and triggered by those unmet needs, an interest in the mechanical properties of the cornea has emerged. Typical examples of mechanical properties are elastic modulus and corneal stiffness.

In this pilot study the investigators will test the ability of a new OCT Vibrography system to determine cornea material parameters. More precisely, the investigators will study the oscillation response in human corneas in-vivo using a stimulus mechanism used to induce vibrations by touching the surface of the cornea. A localized vibration source paired together with phase-sensitive OCT to measure the frequency response function of the human cornea and to analyze the dependency of the frequency response function on age. Additionally the investigators will use Brillouin Microscopy data for computer simulations to validate OCT Vibrography results.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 to 79 years
* Healthy normal subjects with no significant eye disease and no significant refractive errors

Exclusion Criteria:

* Volunteers with implanted intraocular lenses
* Volunteers with LASIK or any other eye surgery, and monocular volunteers
* Volunteers with restricted mobility, who cannot stand up, walk or sit still on a chair without a back
* Subjects who do not or cannot understand the instructions for imaging
* Subjects with diabetes, glaucoma family history
* Subjects who are pregnant and/or breastfeeding.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects to successfully complete OCT Vibrography without serious unanticipated adverse events related to application of the device. | 1 year
  Frequency and severity of all treatment-related adverse events

SECONDARY OUTCOMES:
Validation of OCT Vibrography data by means of Brillouin microscopy measurements of the in-vivo cornea | 1 year
  Use of Brillouin microscopy in-vivo data for computer simulations to validate OCT Vibrography results.

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Hyun Yun, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] de Sanctis U, Loiacono C, Richiardi L, Turco D, Mutani B, Grignolo FM. Sensitivity and specificity of posterior corneal elevation measured by Pentacam in discriminating keratoconus/subclinical keratoconus. Ophthalmology. 2008 Sep;115(9):1534-9. doi: 10.1016/j.ophtha.2008.02.020. Epub 2008 Apr 11. PMID 18405974
- [Background] Li X, Rabinowitz YS, Rasheed K, Yang H. Longitudinal study of the normal eyes in unilateral keratoconus patients. Ophthalmology. 2004 Mar;111(3):440-6. doi: 10.1016/j.ophtha.2003.06.020. PMID 15019316

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03230981/Prot_SAP_000.pdf